CLINICAL TRIAL: NCT04513119
Title: The Short-term Efficacy of Novel No-touch Combined Directional Perfusion Radiofrequency Ablation in the Treatment of Small Hepatocellular Carcinoma With Cirrhosis.
Brief Title: The Short-term Efficacy of Novel NTDP-RFA in the Treatment of Small HCC With Cirrhosis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, fengkai, associate professor, Southwest Hospital, China
Other Study IDs: cstc2019jscx-msxmX0230
Record Dates: First submitted 2020-07-31; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma Stage I; Radiofrequency Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the short-term efficacy of novel no-touch combined directional perfusion radiofrequency ablation in the treatment of small hepatocellular carcinoma with cirrhosis.

DETAILED DESCRIPTION:
Liver cancer is the fourth leading cause of cancer-related deaths globally. Hepatocellular carcinoma (HCC) accounts for 70% to 85% of primary HCC and is the leading cause of death in patients with cirrhosis. We developed a novel no-touch combined directional perfusion radiofrequency ablation system.By inserting two or more electrodes around the tumor and activating them simultaneously.The hypertonic saline solution can be directed into the focal tissue from a lateral pore through a tube within the electrode to provide more uniform and thorough necrosis.The maximum ablation volume was increased while the loss of normal tissue in the non-injection direction was reduced, thus reducing the incidence of postoperative complications. Therefore, the purpose of this study was to evaluate the short-term efficacy of novel no-touch combined directional perfusion radiofrequency ablation in the treatment of small hepatocellular carcinoma with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Primary hepatocellular carcinoma with a background of cirrhosis
* Single shot with diameter ≤ 3cm
* The tumor did not invade portal vein, hepatic vein trunk and secondary branches
* Child Pugh A/B
* ICG-R15 ≤ 30%
* 18-70 years old
* The follow-up time reached 2 years

Exclusion Criteria:

* The follow-up time is less than 2 years
* multiple lesions or diameter > 3cm
* Previous history of upper gastrointestinal bleeding or severe hypersplenism
* Patients with extrahepatic or lymph node metastasis
* Wish to receive liver transplantation and hepatectomy
* The lesion is adjacent to the gallbladder, important blood vessels and bile ducts in the hilum of the liver and important organs around
* severe bleeding tendency, platelet count < 50 × 10^9/L, or prothrombin time prolonged > 3s
* Other anti-tumor therapies were accepted before surgery

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with primary hepatocellular carcinoma with cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of local tumor progression (LTP) | two-years local tumor progression-free survival
  LTP was defined as the appearance of new tumor foci near 2 cm at the ablative margin after the local eradication of all tumor cells with RFA

SECONDARY OUTCOMES:
Tumor-free survival | two-years tumor-free survival
  The tumor did not recur after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kuansheng Ma, Ph.D, Study Director — Institute of hepatobiliary surgery,Southwest Hospital
Locations (1):
- Institute of hepatobiliary surgery,Southwest Hospital, Chongqing, Chongqing Municipality, China